CLINICAL TRIAL: NCT04232319
Title: Feasibility of a Sleep Hygiene Education Program for Sleep Issues in Breast Cancer Survivors
Brief Title: Feasibility and Effectiveness of a Sleep Hygiene Education Program for Sleep Issues in Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID this study was never started.
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UT BCS Sleep Study
Record Dates: First submitted 2019-11-08; First posted 2020-01-18 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Sleep Hygiene
Keywords: Breast cancer, sleep, intervention; Sleep; Intervention; Self-management
MeSH Terms: conditions — Breast Neoplasms; Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Hygiene Training (Experimental): The intervention will be delivered online by an occupational therapist. The intervention consists of 3 weekly sessions; each session will be 30-45 minutes long. The focus of the intervention is to teach breast cancer survivors sleep hygiene strategies to improve their sleep.
  Interventions: Behavioral: Sleep Hygiene Training

INTERVENTIONS:
Behavioral: Sleep Hygiene Training — The intervention will last approximately 45 minutes, and will be provided once/week for 3 weeks. The intervention is delivered "live" using web-cameras (e.g., Microsoft Zoom).
  Registered and licensed occupational therapists will deliver the intervention. Each week, the interventionist will guide the participant through a workbook to provide knowledge regarding sleep hygiene strategies and examples on how to apply these strategies to improve sleep quality.

SUMMARY:
The proposed research will assess the feasibility and preliminary effectiveness of a Sleep Hygiene Program for Breast Cancer Survivors. Participants will complete assessments related to sleep issues, participate in a Sleep Hygiene Program, and complete another assessment post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with breast cancer and not currently receiving active treatment in the form of chemotherapy or radiation therapy,
2. at least 18 years of age,
3. women
4. score > 5 on the Pittsburgh Sleep Quality Index
5. Participant has a smartphone that operates on the Android or Apple platform
6. Participant is able to use the Ecological Momentary Assessment application in the morning
7. functional English fluency and literacy

Exclusion Criteria:

1. self-reported history of diagnosis of co-morbidities that have been associated with poor sleep and fatigue: chronic insomnia, chronic fatigue syndrome, unstable heart, lung, or neuromuscular disease, insulin-dependent diabetes, sleep apnea, chronic oral steroid therapy, and night-shift employment.
2. Currently taking a pharmacological sleep aide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Quality (Pittsburgh Sleep Quality Index) | Baseline to 7 weeks
  Measures the quality of sleep

SECONDARY OUTCOMES:
Change in Ecological Momentary Assessment of Sleep Quality | Baseline to 7 weeks
  Ecological Momentary Assessments via Smartphone App
Change in Actigraphy-based measure of Sleep | Baseline to 7 weeks
  Actigraphy-based measure of Sleep
Change in knowledge of Sleep Hygiene Strategies (Sleep Hygiene Index) | Baseline to 7 weeks
  Measure individual's knowledge of Sleep Hygiene Strategies
Change in Ecological Momentary Assessment of Sleep Quantity | Baseline to 7 weeks
  Ecological Momentary Assessments via Smartphone App

CONTACTS AND LOCATIONS:
Overall Officials: Ketki D Raina, PhD, OTR/L, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No